CLINICAL TRIAL: NCT06024512
Title: DeepView Snapshot Handheld (DV-H) Comparison Study
Acronym: DHA
Status: Completed | Type: Observational
Sponsor: SpectralMD (Industry)
Responsible Party: Sponsor
Other Study IDs: CLA-PR-03
Record Dates: First submitted 2023-08-24; First posted 2023-09-06 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-08

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Burn — This study is being done to collect pictures of burns using an investigational device called the Spectral MD Deep View Snapshot Handheld (DV-H), similar to a camera. The data collected will be used to assess the performance of the DV-H device, and to determine the device's ability to differentiate healing versus non-healing burn tissue. This device, if approved, is expected to give caregivers a better understanding of what parts of burn wounds will likely not heal on their own and as a tool used by the military in the field. This current study involves the collection of images over the course of your clinical treatment and follow-up according to your routine standard of care. The device will not be used to diagnose or prescribe treatment for your burn.

SUMMARY:
his study is being done to collect pictures of burns using an investigational device called the Spectral MD Deep View Snapshot Handheld (DV-H), similar to a camera. The data collected will be used to assess the performance of the DV-H device, and to determine the device's ability to differentiate healing versus non-healing burn tissue. This device, if approved, is expected to give caregivers a better understanding of what parts of burn wounds will likely not heal on their own and as a tool used by the military in the field. This current study involves the collection of images over the course of your clinical treatment and follow-up according to your routine standard of care. The device will not be used to diagnose or prescribe treatment for your burn

ELIGIBILITY:
Inclusion Criteria:

.Age >18 years and able to give informed consent or have a Legally Authorized Representative (LAR) able to do so;

* Life expectancy > 6 months;
* Thermal burn mechanism (flame, scald, or contact);
* The Study Burn(s) occurred less than 72 hours prior to the time of first imaging;
* Minimum burn wound size for patients is 0.5% TBSA per region
* Have 2 - 4 regions of their clinical burn(s) that meet the criteria for a Study Burn; and

Exclusion Criteria:

* Patients will be excluded if any of the following conditions apply:

  * Burn pattern distribution isolated to head, face, neck, hands, feet, genitalia, and/or joints;
  * Subject has burns involving > 50% total body surface area (TBSA);
  * Sepsis at the time of enrollment determined by diagnosis made by Principal Investigator or Sub-Investigator;
  * Immunosuppression/radiation/chemotherapy < 3 months prior to enrollment;
  * Concurrent use of investigational products with a known effect on the burn sites; and/or
  * Any condition that in the opinion of the Investigator may prevent compliance with the study requirements or compromise subject safety.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The goal of this prospective study is to evaluate Study Burns from up to 22 Subjects. Adult will be defined as Subjects 18 years of age or older.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
DeepView Snapshot Handheld (DV-SSH) Comparison Study Protocol | 3 months
  The primary objective of this study is to demonstrate that the proposed SA-MSI sensor is equivalent or better than the current LC-MSI sensor.
  To conduct this test, we will compare the performance of the burn assessment AI algorithm using the image sensor as input data to the same Algorithm using the lens cluster data as an input.

CONTACTS AND LOCATIONS:
Locations (1):
- LSU Health New Orleans University Medical Center New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is still in motion.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year